CLINICAL TRIAL: NCT04363489
Title: The CEDiD Study (COVID-19 Early Diagnosis in Doctors and Healthcare Workers)
Acronym: CEDiD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CEDiD Study
Record Dates: First submitted 2020-04-23; First posted 2020-04-27 (Actual); Last update posted 2021-03-19 (Actual); Status verified 2020-04

CONDITIONS: Covid19
Keywords: COVID-19; wearable medical devices; data analytics; doctors
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — COVID-19 PCR Swabs
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: Wearable Medical Device (Empatica E4) — A wearable medical device (Empatica E4) which is a smart wristband that detects skin temperature, heart rate and sleep. It is CE and FDA approved.
Diagnostic Test: COVID-19 PCR Swab — COVID-19 PCR Swab will be self-taken by doctors every day. Fischer nasopharyngeal PCR Swabs
Diagnostic Test: Pulse Oximeter — Participants will measure their oxygen saturations every day, and report them on the survey. Pulmolink A310 pulse oximeters

SUMMARY:
This is a prospective observational cohort study of healthcare workers working in high-risk COVID-19 clinical areas, monitoring heart rate, sleep and temperature, correlating with daily self-reported symptoms, oxygen saturations and PCR Swabs. It will provide information about how many healthcare workers develop COVID-19, what their clinical observations and symptoms are.

DETAILED DESCRIPTION:
During the COVID-19 Pandemic, doctors and other healthcare workers who work in COVID+ wards, intensive care unit and the accident and emergency department are at high risk of developing COVID-19 infection.

In April 2020, 14.6% of doctors were off sick with suspected or confirmed COVID-19 infection. Meanwhile, 17.9% of COVID+ patients are thought to be asymptomatic. Therefore, healthcare workers are also high-risk of spreading infection to patients, colleagues and their families.

This is a prospective observational cohort study that leverages wearable medical device technology and data analytics to develop an algorithm for early detection of COVID-19 infection in healthcare workers.

A total of 60 healthy healthcare workers working within high-risk COVID-19 clinical areas will be asked to wear a wearable medical device that measures their heart rate, skin temperature and sleep during non-working hours. They will take daily swabs for COVID-19 from themselves, measure their oxygen levels daily, and answer a survey of self-reported symptoms daily for the 30 day study period.

These will then be analyzed to develop an algorithm for early detection of COVID-19 in healthcare workers, and help to inform future workforce decisions, to promote welfare and prevent the spread of COVID-19.

ELIGIBILITY:
Inclusion Criteria

* Healthy healthcare professionals of any age

Exclusion Criteria

* Previous PCR/Antibody positive test for COVID-19
* Not working in high-risk COVID-19 area (ICU, A&E, COVID positive wards)
* Involved in COVID-19 Vaccine Trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy healthcare workers who work in high-risk COVID-19 areas, and have not themselves had a PCR/Antibody positive diagnosis of COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-08-20 (Actual); Primary Completion 2021-05-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
COVID-19 Infection | 30 days
  Number of Healthcare Workers who have a new PCR positive diagnosis of COVID-19

SECONDARY OUTCOMES:
Symptoms | 30 days
  What new symptoms healthcare workers develop when they develop COVID-19 infection
Clinical Observations | 30 days
  What healthcare workers observations are when they develop COVID-19 infection including: Oxygen saturations, Heart Rate, Skin Temperature

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Zargaran, MBBS, Study Director — King's College London / Guy's and St Thomas' NHS Foundation Trust; Anne Greenough, Study Chair — King's College London; Dina Radenkovic, MBBS, Study Director — King's College London / Guy's and St Thomas' NHS Foundation Trust; Rocio Martinez-Nunez, PhD, Study Director — King's College London; Kariem El-Boghdadly, Principal Investigator — Guy's and St Thomas' NHS Foundation Trust
Locations (1):
- Guy's and St Thomas' NHS Foundation Trust, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Zargaran A, Sousi S, Colville G, Radcliffe G, Malek R, Douiri A, El-Boghdadly K, Nebbia G, Martinez Nunez RT, Greenough A. COVID-19 Early Detection in Doctors and Healthcare Workers (CEDiD) study: a cohort study on the feasibility of wearable devices. BMJ Open. 2025 Apr 5;15(4):e089598. doi: 10.1136/bmjopen-2024-089598. PMID 40187781